CLINICAL TRIAL: NCT01004653
Title: An Open-Label Clinical Trial With Split-virion Influenza A/H1N1 Vaccines in Healthy Elders
Brief Title: A Clinical Trial of Split-virion Influenza A/H1N1 Vaccines
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sinovac Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PRO-PanFlu-4001-1
Record Dates: First submitted 2009-10-29; First posted 2009-10-30 (Estimated); Last update posted 2013-03-15 (Estimated); Status verified 2013-03

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

ARMS (1):
- H1N1 influenza A Vaccine (Split virion), Inactivated (Experimental): 15 μg H1N1 influenza A Vaccine (Split virion), Inactivated
  Interventions: Biological: H1N1 influenza A Vaccine (Split virion), Inactivated

INTERVENTIONS:
Biological: H1N1 influenza A Vaccine (Split virion), Inactivated — 100 elders were assigned to receive one dose of 15μg H1N1 influenza A Vaccine (Split virion), Inactivated

SUMMARY:
A single center, Open-Label phase IV clinical trial is to be conducted in healthy elders (equal to or more than 61 years to evaluate the immunogenicity and safety of Sinovac's 15μg H1N1 influenza A Vaccine (Split virion), Inactivated.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female aged 60 and older
2. Be able to show legal identity card for the sake of recruitment
3. Volunteers are able to understand and sign the informed consent

Exclusion Criteria:

1. Cases, cured cases and close contact of influenza A (H1N1) virus
2. Women of pregnancy, lactation or about to be pregnant in 60 days
3. Subject that has a medical history of any of the following: allergic history, or allergic to any ingredient of vaccine, such as egg, egg protein, etc
4. Serious adverse reactions to vaccines such as anaphylaxis, hives, respiratory difficulty, angioedema, or abdominal pain
5. Autoimmune disease or immunodeficiency
6. Asthma that is unstable or required emergent care, hospitalization or intubation during the past two years or that required the use of oral or intravenous corticosteroids
7. Diabetes mellitus (type I or II), with the exception of gestational diabetes
8. History of thyroidectomy or thyroid disease that required medication within the past 12 months
9. Serious angioedema episodes within the previous 3 years or requiring medication in the previous two years
10. Bleeding disorder diagnosed by a doctor (e.g. factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties with IM injections or blood draws
11. Active malignancy or treated malignancy for which there is not reasonable assurance of sustained cure or malignancy that is likely to recur during the period of study
12. Seizure disorder other than:

    * Febrile seizures under the age of two years old
    * Seizures secondary to alcohol withdrawal more than 3 years ago, or
    * A singular seizure not requiring treatment within the last 3 years
13. Asplenia, functional asplenia or any condition resulting in the absence or removal o the spleen
14. Guillain-Barre Syndrome
15. Any history of immunosuppressive medications or cytotoxic medications or inhaled corticosteroids within the past six months (with the exception of corticosteroid nasal spray for allergic rhinitis or topical corticosteroids for an acute uncomplicated dermatitis)
16. History of any blood products or seasonal influenza vaccine administration within 3 months before the dosing
17. Administration of any other investigational research agents within 30 days before the dosing
18. Administration of any live attenuated vaccine within 30 days before the dosing
19. Administration of subunit or inactivated vaccines, e.g., pneumococcal vaccine, or allergy treatment with antigen injections, within 14 days before the dosing
20. Be receiving anti-TB prophylaxis or therapy currently
21. Axillary temperature > 37.0 centigrade at the time of dosing
22. Psychiatric condition that precludes compliance with the protocol:

    * Past or present psychoses
    * Past or present bipolar disorder requiring therapy that has not been well controlled on medication for the past two years
    * Disorder requiring lithium
    * Suicidal ideation occurring within five years prior to enrollment
23. Any medical, psychiatric, social condition, occupational reason or other responsibility that, in the judgment of the investigator, is a contraindication to protocol participation or impairs a volunteer's ability to give informed consent

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-09; Primary Completion 2009-10 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Evaluate immunogenicity of split-virion influenza A （H1N1）vaccine in elders | Sep. 2009- Oct. 2009

SECONDARY OUTCOMES:
Evaluate Safety of split-virion influenza A （H1N1）vaccine in elders | Sep. 2009- Oct. 2009

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Centers for Diseases Control and Prevention, Beijing, China